CLINICAL TRIAL: NCT05896085
Title: Game Based Assessment of Emotion-regulation Skills in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D of Clinical Psychology, Babes-Bolyai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REThin Academy - assessment
Record Dates: First submitted 2023-05-26; First posted 2023-06-09 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Assessment; Emotion Regulation
Keywords: online therapeutic game; emotion regulation; college students; mental health; game-based assessment
MeSH Terms: conditions — Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- REThink game (Experimental): Participants will complete the online standardized scales and then complete the REThink therapeutic game's assessment system in 3D or VR version.
  Interventions: Other: REThink game

INTERVENTIONS:
Other: REThink game — The Rethink therapeutic game is an online game developed based on Rational-Emotive Behavioral Therapy and has two versions: for children and adolescents and for adults. The Rethink therapeutic game for adults is available in 3D and VR version and consists of four levels, each of them training a specific emotion regulation ability such as: emotional awareness, mindfulness, cognitive change

SUMMARY:
The aim of this study will be to investigate the validity of the in-game performance measurements or scores as indicators of students'ER abilities.

ELIGIBILITY:
Inclusion Criteria:

* first year student at Babes-Bolyai University
* internet and PC access to complete the scales and game

Exclusion Criteria:

* no internet or PC access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Mental Health | baseline, pre-intervention
  The General Health Questionnaire, 12-item version (GHQ-12 by Goldberg &Williams,1988 is a self-report scale measuring mental health on a 6-point Likert scale ranging from 0 "never" to 5 "everyday" where grater scores represents better mental health.
Emotion regulation | baseline, pre-intervention
  The Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski, Kraaij, & Spinhoven, 2001) is a self-report scale measuring emotion regulation on a 5 point Likert scale ranging from "almost never" to "almost always". It had 9 subscales representing 9 emotion regulation strategies and grater scores represents grater involvement in using that strategy.

SECONDARY OUTCOMES:
MAAS | baseline, pre-intervention
  Brown, K. W., & Ryan, R. M. (2003). Mindful attention awareness scale. Journal of personality and social psychology The Mindfull Attention Awareness Scale is a 15 items self-report scale, rated on 5 point Likert scale from "almost never" to "almost always", where greater scores represents better mindfulness.
Rational and irrational cognition | baseline, pre-intervention
  Attitudes and Beliefs Scale 2 Abbreviated Version (ABS-2 - AV; Hyland et al. 2014) is a 24-items self-report scale that measures the presence of rational and irrational cognitions. It has two subscales one for rational cognitions and one for irrational cognitions. Greater scores at each scale represents more rational/irrational cognitions in an individual. Items are rated on a 5 point Liker scale ranging from "totally disagree" to "totally agree".
Atention to positive and negative information | baseline, pre-intervention
  Attention to Positive and Negative Information Scale Noguchi, K., Gohm, C. L., & Dalsky, D. J. (2006). Cognitive tendencies of focusing on positive and negative information. Journal of Research in Personality, 40(6), 891-910. It is a self- report scale for measuring the attention to positive or negative information. It is rated on a 5 point Likert scale ranging "not at all" to " completely conform"and it has 29 items. Grater scores at this scale represent more attantion toward a specific type of information-negative or positive.
emotional distress | baseline, pre-intervention
  Distress and positive emotions: Profile of Affective Distress Plus; PED Opris & Macavei, 2007 is a self-report scale that measure distress. It had 42 items rated on a 5 point Liker scale ranging from "not al all" to "a lot" and grater scores represent grated level of distress.
emotional awareness | baseline, pre-intervention
  The Emotion Awareness Questionnaire (EAQ, Rieffe et al., 2008) is a 32-item questionnaire on a three-point Liker scale, from 0 "not true" to 2 "certainly true" where greater scores represents better levels of emotional awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No